CLINICAL TRIAL: NCT01772459
Title: Internet-administered Adolescent Scoliosis Questionnaires Compared With Traditional Pencil and Paper Versions: a Randomized Crossover Design
Brief Title: Paper vs. Internet
Acronym: P vs I
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: iACT - Innovations in Acute Care and Technology (Unknown)
Responsible Party: Sponsor
Other Study IDs: H10-01785; CW10-0184 (Other: UBC C&W Research Ethics Board)
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Idiopathic Scoliosis; Adolescent
Keywords: Scoliosis; Adolescents; Questionnaire; Reliability
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Paper/Paper: This group will complete paper questionnaires at baseline and two week follow up.
- Paper/Internet: This group will complete paper questionnaires at baseline and internet questionnaires at two week follow up.
- Internet/Paper: This group will complete internet questionnaires at baseline and paper questionnaires at two week follow up.
- Internet/Internet: This group will complete internet questionnaires at baseline and two week follow up.

SUMMARY:
Research has shown that questionnaires completed on the internet have the potential to provide more complete and honest data with fewer errors in a more efficient manner than questionnaires completed using the paper and pencil format. Despite the numerous advantages of internet-administered questionnaires, it is important to make sure that the internet questionnaires will yield comparable results to the well-established paper and pencil versions. No one has studied internet administration of scoliosis specific questionnaires in adolescents with scoliosis. The investigators will test whether the internet administration of scoliosis questionnaires is as reliable as the traditional paper and pencil version. The investigators predict that the internet-administered questionnaire will provide the same reliability as the paper-administered questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Aged 10-18
* Male or female
* Diagnosis of Adolescent or Juvenile Idiopathic Scoliosis
* Home access to computer and internet
* Capable or oral and written communication in English

Exclusion Criteria:

* Unable to communicate in English

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents with idiopathic scoliosis will be asked to participate during visits to the orthopaedic spine clinic at BC Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2010-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
To test the reliability of the internet-administered PODCI and SRS-30 questionnaires in adolescents with idiopathic scoliosis | 2 weeks
  The reliability of internet-administered questionnaires will be determined by comparison to standard paper questionnaire implementation.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Reilly, MD, FRCSC, Principal Investigator — University of British Columbia
Locations (1):
- British Columbia Children's Hospital, Vancouver, British Columbia, Canada